CLINICAL TRIAL: NCT00178074
Title: The Effects of Sleep Deprivation on Antidepressant Response in Geriatric Depression: Neurometabolic Substrates Studied With PET
Brief Title: The Effects of Sleep Deprivation on Antidepressant Response
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: R01MH037869-03 (NIH); 980753; DATR A4-GPS
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Unipolar Depression
Keywords: depression; imaging; PET; elderly; late life; sleep deprivation
MeSH Terms: conditions — Depressive Disorder; Depression; Sleep Deprivation | interventions — Magnetic Resonance Spectroscopy

INTERVENTIONS:
Behavioral: total sleep deprivation
Procedure: PET imaging

SUMMARY:
This study will use positron emission tomography (PET) to examine the effect of sleep deprivation on brain function.

DETAILED DESCRIPTION:
This study seeks to better understand the effect of sleep deprivation (TSD) on brain function using Positron Emission Tomography (PET). PET is an established research procedure that produces images of the brain. The purpose of these images is to show changes in brain activity associated with sleep deprivation. The neurochemical mechanisms underlying the TSD acceleration of antidepressant efficacy have not been identified. An understanding of these neurochemical processes may lead to the development of pharmacologic strategies that would accelerate antidepressant response or more directly to the development of antidepressant treatments that are more efficacious.

This study will be conducted in collaboration with Dr. Charles Reynolds' ongoing protocol "Geriatric Depression: Neurobiology of Treatment" (IRB #970356). The impetus for the clinical studies is the finding that the clinical response to antidepressant treatment in geriatric depressed patients is delayed, with the median time to remission reported as up to 12 weeks. Thus, the development of a strategy to accelerate treatment response would represent a substantial contribution to the treatment of geriatric depression. One approach that has been reported to accelerate antidepressant response in mid-life depression is one night of total sleep deprivation (TSD) prior to initiating antidepressant treatment. TSD has also been shown to improve mood in depressed patients, the response to TSD may distinguish subsequent treatment responders from non-responders and depressive relapse may occur after naps or a night of recovery sleep. The neurochemical mechanisms underlying the TSD acceleration of antidepressant efficacy have not been identified. An understanding of these neurochemical processes may lead to the development of pharmacologic strategies that would accelerate antidepressant response or more directly to the development of antidepressant treatments that are more efficacious.

Advancements in brain imaging technology and radiotracer chemistry have made it possible to measure metabolic activity and specific neurochemical mechanisms using Positron Emission Tomography (PET). The proposed studies represent the initial step in characterizing the neurochemical alterations produced by TSD and the impact of TSD on antidepressant response by TSD in geriatric depressed patients using PET and a radiotracer for brain glucose metabolism, [18F]-2deoxy-2-fluoro-D-glucose ([18F]-2DG). Having established the regional metabolic alterations associated with sleep deprivation and recovery sleep in patients who are subsequent treatment responders and compared the metabolic changes with treatment non-responders, future studies will be undertaken using neuroreceptor radiotracers to define the specific neurochemical pathways subserving the regional pattern of metabolic alterations. The glucose metabolic response to sleep deprivation in mid-life depression has been investigated at the UPMC PET Facility and at other institutions (e.g. Dube et al., in preparation, Wu et al., 1991, 1992). The studies performed in the geriatric depressed patients will be compared with the PET studies conducted in mid-life depressed patients to assess the contribution of the aging process to the neurometabolic response to sleep.

For information on related studies, please follow these links:

http://clinicaltrials.gov/show/NCT00177294

http://clinicaltrials.gov/show/NCT00178035

ELIGIBILITY:
Inclusion Criteria:

Patients:

* DSM-IV criteria for current major depressive disorder
* Score of 15 or higher on the HRSD (17 item)
* Score of 17 or higher on the Folstein Mini-Mental Status Exam

Control Subjects:

-No history of psychiatric disorder or neurological illness

Exclusion Criteria:

Patients:

* lifetime diagnosis of any psychotic disorder
* bipolar disorder
* alcohol or drug abuse within the last 6 months
* No contraindication to SSRI therapy
* History of seizure disorder

Both Patient and Control Subjects:

-Current diagnosis of diabetes or significantly altered plasma glucose levels

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 1999-02; Study Completion 2003-04

PRIMARY OUTCOMES:
To gain an understanding of the neurochemical processes that may lead to development of pharmacologic strategies that would accelerate antidepressant response or more directly to the development of antidepressant treatments.
PET study
Regional glucose metabolic rates and regional [18F]-altanserin binding
MRI scan

SECONDARY OUTCOMES:
Beck Depression Inventory
Profile of Mood States
Serum anticholinergicity and paroxetine blood levels
SCID
Hamilton Depression Rating Scale
Folstein Mini-Mental State Exam

CONTACTS AND LOCATIONS:
Overall Officials: Charles F Reynolds III, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States